CLINICAL TRIAL: NCT00365183
Title: Phase II Trial of Motexafin Gadolinium and Pemetrexed (Alimta®) for Second Line Treatment in Patients With Non-Small Cell Lung Cancer
Brief Title: Trial of Motexafin Gadolinium and Pemetrexed (Alimta®) for Second Line Treatment in Patients With Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0228
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Non-Small Cell Lung Carcinoma
Keywords: Non Small Cell Lung Cancer; Lung Cancer; Metastatic Lung Cancer; Inoperable Lung Cancer; Advanced Lung Cancer; Large Cell Lung Cancer; Adenocarcinoma, lung; Squamous Cell Carcinoma, lung; Squamous Cell Lung Cancer; Large Cell Carcinoma, lung; Cancer of the Lung; Carcinoma; Bronchogenic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Squamous Cell; Carcinoma, Large Cell; Carcinoma | interventions — motexafin gadolinium; Pemetrexed

ARMS (1):
- Xcytrin® (motexafin gadolinium) (Experimental)
  Interventions: Drug: Motexafin gadolinium and pemetrexed

INTERVENTIONS:
Drug: Motexafin gadolinium and pemetrexed — 1 dose of MGd 15 mg/kg and pemetrexed 500 mg/m2 once during the first week of every 3-week treatment cycle for a maximum of 12 cycles
  Other Names: MGd and Alimta®

SUMMARY:
The goals of this study are:

* to determine if the combination of two drugs, motexafin gadolinium and pemetrexed, may be an effective treatment for patients with non-small cell lung cancer (NSCLC) who have had one previous chemotherapy regimen that included a platinum containing drug such as cisplatin or carboplatin.
* to assess response to treatment in patients with NSCLC six months after beginning study treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Stage IIIb, metastatic, or recurrent NSCLC patients who have received one prior platinum-based chemotherapy regimen
* ECOG performance status score of 0 or 1

Exclusion Criteria:

* Laboratory values indicating inadequate function of bone marrow, liver, or kidneys
* Symptomatic or uncontrolled brain metastases
* Evidence of meningeal metastasis
* > 1 prior regimen (not counting adjuvant or neo-adjuvant cytotoxic chemotherapy if completed > 12 months prior to regiment)
* Medical condition that would increase risk if treated with motexafin gadolinium or impair ability to complete study procedures and assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
6 month progression free survival | up to 2 years
  proportion of patients who are still alive and who have not progressed clinically or radiographically 6 months after receiving their first dose of MGd.

SECONDARY OUTCOMES:
Time to disease progression | up to 2 years
  Time to progression is defined as the time from first dose of MGd to first evidence of progression.
Overall survival | up to 2 years
  Patient population for this endpoint consists of all patients receiving at least 1 dose of MGd and pemetrexed.
Progression free survival | up to 2 years
  Progression-free survival is defined as the time from first dose MGd to the earlier of progression or death.
Response rate (CR+PR) by RECIST criteria | up to 2 years
  Patient population for this endpoint consists of all patients receiving at least 1 dose of MGd and pemetrexed and underwent at least response assessment.
Duaration of reponse (CR+PR) | up to 2 years
  Duration of response (CR + PR) is defined as the time from first response to the time of disease progression.
Clinical benefit rate (CR+PR+SD) | up to 2 years
  Patient population for this endpoint consists of all patients receiving at least 1 dose of MGd and pemetrexed and underwent at least response assessment
Safety and tolerability of MGd and pemetrexed | up to 2 years
  All patients who receive any MGd will be included in the safety summaries and analyses

CONTACTS AND LOCATIONS:
Overall Officials: Martin Edelman, MD, Study Chair — University of Maryland, Greenbaum Cancer Center
Locations (11):
- United States (11):
  - Huntington Beach, California
  - Long Beach, California
  - Chicago, Illinois
  - Baltimore, Maryland
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Santa Fe, New Mexico
  - Armonk, New York
  - Columbus, Ohio
  - Seattle, Washington

REFERENCES:
- [Background] Biaglow JE, Miller RA. The thioredoxin reductase/thioredoxin system: novel redox targets for cancer therapy. Cancer Biol Ther. 2005 Jan;4(1):6-13. doi: 10.4161/cbt.4.1.1434. Epub 2004 Jan 8. PMID 15684606
- [Background] Evens AM. Motexafin gadolinium: a redox-active tumor selective agent for the treatment of cancer. Curr Opin Oncol. 2004 Nov;16(6):576-80. doi: 10.1097/01.cco.0000142073.29850.98. PMID 15627019